CLINICAL TRIAL: NCT01601093
Title: Phase Ⅱ Study on Ceftazidime Sodium and Sulbactam Sodium for Injection(2:1) for Treatment of Respiratory and Urinary System Infection
Brief Title: Study on Ceftazidime and Sulbactam Sodium for Injection (2:1) for Treatment of Respiratory and Urinary Tract Infection
Acronym: CAZ-SBT
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: other project got priority
Sponsor: Xiangbei Welman Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2008L03354
Record Dates: First submitted 2012-04-27; First posted 2012-05-17 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Tract Infections; Urinary Tract Infections
Keywords: Respiratory and urinary tract infections; Ceftazidime and Sulbactam Sodium for Injection (2:1); Phase Ⅱ
MeSH Terms: conditions — Respiratory Tract Infections; Urinary Tract Infections | interventions — Population Groups; Contraceptives, Oral; Cefoperazone; Sulbactam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose (Experimental): Ceftazidime 3g
  Interventions: Drug: High dose
- Low dose (Experimental): Ceftazidime 2g
  Interventions: Drug: Low dose
- CFP/SUB (Active Comparator): Cefoperazone and sulbactam sodium for injection(2:1)
  Interventions: Drug: Cefoperazone and Sulbactam Sodium (CFP/SUB)

INTERVENTIONS:
Drug: High dose — Ceftazidime 3g, iv, bid and Sulbactam Sodium 1.5g, iv, bid for 5-14days.
  Other Names: high dose group
  Arms: High dose
Drug: Low dose — Ceftazidime 2g, iv, bid and Sulbactam Sodium 1g, iv, bid for 5-14days.
  Arms: Low dose
Drug: Cefoperazone and Sulbactam Sodium (CFP/SUB) — Cefoperazone 2g, iv, bid and Sulbactam Sodium 1g, iv, bid for 5-14days.
  Other Names: CFP/SUB(2:1)
  Arms: CFP/SUB

SUMMARY:
In the proposed study, the investigators plan to evaluate the efficacy and safety of Ceftazidime Sodium and Sulbactam Sodium for Injection(2:1) for the treatment of respiratory and urinary tract acute bacterial infection.

DETAILED DESCRIPTION:
Ceftazidime is a third-generation cephalosporins. Ceftazidime sodium and sulbactam sodium for injection (2:1)plays a therapeutic role by the former inhibiting bacterial cell wall synthesis，the latter making irreversible competitive inhibition of β-lactamase.The antimicrobial effect of ceftazidime can be enhanced by the two combined. The compound specifically aims to the mechanism of bacterial resistance, extending the life of ceftazidime in the treatment-resistant pathogen infections.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who qualify for moderate and severe acute respiratory or urinary tract bacterial infection of acute bacterial infections need for systemic antibiotic therapy.
2. Hospital patients or good compliance clinic patients, who were more than 18 years old and less than 70 years old, Gender: both.
3. Patients who do not take other antibiotic medications before screening period.
4. Patients who have no severe liver, kidney and hematopoietic system of diseases (Both AST and ALT are less than 1.5 times of the upper limit of normal and Cr is in normal range)
5. Pathogenic bacteria was resistant to ceftazidime and sensitive to both of test drugs and contrast drugs.
6. Women of childbearing was to be negative pregnancy test and agree to take contraceptive measures during the trial.
7. Patients were volunteers and signed informed consent from.

Exclusion Criteria:

1. Patients were hypersusceptibility to the test drug or other penicillins ,β-lactamase inhibitor
2. Pathogenic bacteria was sensitive to ceftazidime or resistant to ceftazidime,test drugs and control drugs.
3. Patients who need to take other antibiotic medicine because of concurrent infection.
4. Patients who took medicine which affected efficacy evaluations and safety evaluations such as aspirin, indomethacin, phenylbutazone, sulfanilamide, disulfiram and probenecid in the trial.
5. Patients who took risks of severe drug interactions because of drug combination.
6. Patients who were complicated by other diseases and thought to affect efficacy evaluations or poor compliance.
7. Pregnant and Lactating women
8. Drug addicts and alcoholics.
9. Patients who once was selected in this trial.
10. Patients who participated in other clinical trials in the past three months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2011-11; Primary Completion 2022-08-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
The rate of bacterial clearance | two years
  end of treatment of bacteriological efficacy(bactercial clearance) The fore-and-aft changes of clinical symptoms and signs after discontinuation of durgs

SECONDARY OUTCOMES:
Number of participants with Adverse Events | two years
  the incidence(%)of allergies, skin rashes, shock,death, etc.

CONTACTS AND LOCATIONS:
Overall Officials: hong wh wang, doctor, Principal Investigator — The first affliated hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital With Medical University, Nanjing, Jiangsu, China